CLINICAL TRIAL: NCT02471170
Title: Protocol to Permit the Acquisition of Circulating Tumor Material in Pancreatic Diseases
Status: Enrolling by invitation | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 02215
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Diseases
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The frequency of research blood collection will not exceed 60 mL in a 1 week period and will not occur more frequently than 4 times in an 8 week period.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to collect blood samples to detect potential markers of pancreatic cancer in the blood and link these findings to medical and health information. Information from this study may help to provide insight into the detection of pancreas cancer in the blood before it can be found by other methods or provide a method of monitoring the status of pancreatic cancer throughout a treatment course. Another purpose of this study is to collect blood to create a biobank.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be a patient at the Hospital of the University of Pennsylvania

   * The subject must be under evaluation and/or treatment for a pancreatic disease
   * The subject must be under evaluation and/or treatment for a non-pancreatic disease. For example, patients undergoing routine colonoscopy within the clinical practice will be asked to consent to provide control samples.
2. The subject must be able to provide informed consent or have an acceptable surrogate capable of giving consent on the subject's behalf
3. The subject must be 18 years of age or older

Exclusion Criteria:

1. The subject or acceptable surrogate does not provide informed consent
2. Subject is a prisoner
3. Subject is under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with pancreatic diseases
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-09-10 (Actual); Primary Completion 2035-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Collection of blood and tissue samples from subjects with pancreatic diseases | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Dwyer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States